CLINICAL TRIAL: NCT05654168
Title: Muscular Morphological Ultrasound Epidemiological Study in Dance Professionals
Acronym: DancersMUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Miguel Ángel Alcocer Ojeda, Master's degree Physiotherapy degree PhD candidate, Universidad de Murcia
Other Study IDs: Task BIBDIG-6394
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Femoracetabular Impingement
Keywords: Dancing; Groin; Pain; Ultrasonography
MeSH Terms: conditions — Femoracetabular Impingement; Pain | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Professional dancers: Professional dancers with and without groin pain
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — The thickness of the musculature to be studied will be measured with ultrasonography

SUMMARY:
This research will determine the presence of groin pain in professional dancers, through a specific questionnaire on the hip joint. Two groups will be formed made up of dancers over 18 years of age, men and women; one with groin pain and one without groin pain. All participants will undergo a functional muscle ultrasound study, where the thickness of the abdominal muscles, lumbar multifidus and gluteus medius and minor will be evaluated, and the relationship between ultrasound neuromuscular changes and groin pain will be verified

DETAILED DESCRIPTION:
The objective of the study is to shed light on the to the complexity of the Diagnosis that Groin Pain (GP) encloses, it is proposed to evaluate with Functional Muscular Ultrasonography Rehabilitative Ultrasound Imaging (RUSI), the layer thickness of the gluteal musculature of the hip and the abdominal and lumbar muscles on a sample of professional dancers over 18 years of age with GP to check if there are differences with professional dancers without GP.

Expected goals:

1. Identify the presence of GP in professional dancers.
2. To compare the ultrasound characteristics of the neuromuscular system between a sample of dancers with GP and a sample of dancers no GP.
3. Verify the relationship between ultrasound neuromuscular changes with GP.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer Professional dancers 18 years or older, and no maximum age limits

Exclusion Criteria:

* Not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • Professional dancers of the National Ballet of Spain
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
RUSI. (REHABILITATIVE ULTRASOUND IMAGING) | Five months
  Taking measurements of the layer thickness of abdominal, lumbar and gluteal muscle groups will be performed, with Toshiba's Nemio XG equipment using a multifrequency convex probe from 3 to 6 MGz.

SECONDARY OUTCOMES:
HAGOS questionnaire | Five months
  Correlate the HAGOS questionnaire with the thicknesses of layer of the different muscle groups analyzed at rest and in contraction in the group with Groin Pain and in the group without Groin pain.

OTHER OUTCOMES:
One- Way ANCOVA | Five months
  One-way ANCOVA will used to compare quantitative muscle ultrasound (QMUS) variables in hip with or without groin pain, controlling for effects of clinical covariates Regression models will used to study the relationship between time of evolution (and if necessary, logarithmic transform will applied to this variable to correct the absence of a normal distribution) as independent variable and the QMUS parameters as dependent variables

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL ANGEL ALCOCER OJEDA, MSc PT, Principal Investigator — Universidad de Murcia; ANTONIA GOMEZ CONESA, PhD, PT, Study Director — Universidad de Murcia
Locations (1):
- Miguel Angel Alcocer Ojeda, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No